CLINICAL TRIAL: NCT06242899
Title: Effects of Short Moderate-intensity Continuous Training With Different Durations on Sedentary Women's Functional Capacity and Physical Activity Enjoyment. A Randomized Clinical Trial.
Brief Title: Short Moderate-intensity Continuous Training on Sedentary Women's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Elena Marques-Sule, Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AL-jouf University036
Record Dates: First submitted 2024-01-23; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 8-minutes short exercise group (Experimental): Participants performed an intervention for 3 sessions/week, over 3 weeks and a cycle ergometer was used. The workout regimen consisted of a structured warm-up lasting 2 minutes. The main exercise phase comprised an 8-minute cycling session performed at 75% of HRmax. Finally, a cool down phase lasting 2 minutes.
  Interventions: Other: Exercise
- 10-minutes short exercise group (Experimental): Participants performed an intervention for 3 sessions/week, over 3 weeks and a cycle ergometer was used. The workout regimen consisted of a structured warm-up lasting 2 minutes. The main exercise phase comprised an 10-minute cycling session performed at 75% of HRmax. Finally, a cool down phase lasting 2 minutes.
  Interventions: Other: Exercise
- 15-minutes short exercise group (Experimental): Participants performed an intervention for 3 sessions/week, over 3 weeks and a cycle ergometer was used. The workout regimen consisted of a structured warm-up lasting 2 minutes. The main exercise phase comprised an 15-minute cycling session performed at 75% of HRmax. Finally, a cool down phase lasting 2 minutes.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise with a cycle ergometer in three phases:
  * Warm-up: the exercise intensity was determined at 50-60% of HRmax obtained in the effort test, and lasted 2 minutes.
  * Short exercise at moderate intensity for 8, 10 or 15 minutes according to group allocation. The exercise was cycling at 75% HRmax determined with an effort test.
  * Cool down: the exercise intensity was determined at 50-60% of HRmax obtained in the effort test, and lasted 2 minutes.

SUMMARY:
Purpose: To determine the effects of three Short Moderate Intensity Continuous Training (SMICT) exercise programs with different durations, on functional capacity, resting heart rate (RHR) and physical activity enjoyment in sedentary women.

Methods: A randomized clinical trial was performed. 45 sedentary women were randomly allocated to either a: i) 8-minutes short exercise group; ii) 10-minutes short exercise group; and iii) 15-minutes short exercise group. All three groups received a short exercise training program at moderate intensity for 3 sessions/week, over 3 weeks. Before and after the interventions, functional capacity was evaluated through the 6-minute walking test, and RHR with a pulse oximeter. Physical activity enjoyment was measured with the Physical Activity Enjoyment Scale after the intervention.

DETAILED DESCRIPTION:
Sedentary lifestyles contribute to 3.2 million annual deaths globally, correlating with increased risks of cardiovascular diseases, obesity, and certain cancers. With women showing notably low physical activity rates, implementing tailored exercise interventions becomes crucial to enhance their activity levels and functionality, potentially mitigating risks associated with high resting heart rates linked to increased mortality, particularly from cardiovascular causes.

This was a randomized clinical trial involving 45 sedentary women split into three groups: 8-minute, 10-minute, and 15-minute exercise durations. All groups underwent moderate-intensity short exercise programs, differing only in duration. Functional capacity (measured by the 6-minute walking test) and resting heart rate (RHR) were assessed at baseline and after the 3-week intervention. Physical activity enjoyment was measured at the intervention's end.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Must be not regularly physically active for more than one month.
* Must be between 18 and 25 years of age.
* Must present a body mass index (BMI) between 18.5-24.9 kg/m2.

Exclusion Criteria:

* BMI≥25 kg/m2.
* Suffer from musculoskeletal or neurological diseases.
* Women with precarious medical conditions.
* Use of medications.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Sedentary women
Enrollment: 45 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Functional capacity | Up to 3 weeks
  6-minutes walking test (6MWT). This test consists of calculating the distance covered by the participant who was instructed to walk as quickly as possible along a 30-meter hallway without running for six minutes. Greater number of meters covered, better functional capacity.
Resting heart rate | Up to 3 weeks
  Resting heart rate was measured with a pulse oximeter. The normal values for oxygen saturation (SpO2) in healthy adults measured by a pulse oximeter are 95% to 100%
Physical activity enjoyment | Up to 3 weeks
  Physical activity enjoyment was measured with a modified version of the Physical Activity Enjoyment Scale (PACES). The scale is comprised of 17 items that are assessed using a 7-point bipolar scale. The final enjoyment score is calculated, and possible scores range from 17 (representing not enjoyable) to 68 (indicating neutral) to 119 (reflecting enjoyable). The higher score indicates greater enjoyment.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Marqués Sulé, PhD, Principal Investigator — Univeristy of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Pines A. Sedentary women: sit less, live more! Climacteric. 2015;18(6):770-2. doi: 10.3109/13697137.2015.1038512. Epub 2015 Apr 14. PMID 25868822